CLINICAL TRIAL: NCT05834673
Title: AtheroSclerotic Cardiovascular disEase Risk assessmenT and treAtment In AustraliaN Primary Care (VICTORION-ASCERTAIN: Implementation Study)
Brief Title: VICTORION-ASCERTAIN: Implementation Study (v-ASCERTAIN)
Acronym: v-ASCERTAIN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Loss of strategic interest by the funding party. The participants' recruitment rate failed to meet the target within the pre-specified recruitment windows.
Sponsor: Monash University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Stephen Nicholls, Program Director of MonashHeart, Intensive Care and Victorian Heart Hospital, Monash University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CKJX839A1AU03R
Record Dates: First submitted 2023-02-20; First posted 2023-04-28 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Atherosclerotic Cardiovascular Disease (ASCVD); Coronary Heart Disease (CHD); Cerebrovascular Disease; Peripheral Arterial Disease (PAD)
Keywords: Hyperlipidaemia; Atherosclerotic Cardiovascular Disease (ASCVD); Hypercholesterolaemia; Lipid lowering therapies; Secondary Cardiovascular Prevention; New Model of Care; Nurse-Led Support Calls; Guideline Directed Management therapy (GDMT); The European Society of Cardiology (ESC) Guidelines
MeSH Terms: conditions — Atherosclerosis; Coronary Disease; Cerebrovascular Disorders; Peripheral Arterial Disease; Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Model (Other): Usual care arm :
  The GPs will be educated on the ESC guidelines and Guideline Directed Management therapy (GDMT) Inclisiran is available for this arm
  Interventions: Other: GP Education
- New Model of Care (Other): Model of care arm The GPs will be educated on the ESC guidelines and Guideline Directed Management therapy (GDMT) The Participants enrolled via these sites arm will be getting receive monthly SMS messages with regards to regarding cardiovascular health and appointment reminders (low touch engagement nudges) In addition, Participants will receive telephone-based support calls from a study nurse trained in motivational interviewing. These telephone calls will cover diet, exercise, medication, and where necessary smoking cessation. A summary of any recommendations will then be sent to the primary care physician via email or letter.
  Inclisiran is available for this arm.
  Interventions: Other: SMS messages; Other: Telephone-based support calls; Other: GP Education

INTERVENTIONS:
Other: SMS messages — Participants will receive monthly SMS messages regarding cardiovascular health (low touch engagement nudges)
  Other Names: Monthly Text Messages
  Arms: New Model of Care
Other: Telephone-based support calls — Participants will receive telephone-based support calls from a study nurse trained in motivational interviewing. These telephone calls will cover diet, exercise, medication, and where necessary smoking cessation. A summary of any recommendations will then be sent to the primary care physician via email or letter.
  Other Names: Nurse Support Calls
  Arms: New Model of Care
Other: GP Education — Education of GPs on the European Society of Cardiology (ESC) guidelines and Guideline Directed Management Therapy

SUMMARY:
The goal of this study is to understand and compare an alternative model of care in comparison to the usual model of care in include male and female participants ≥18 years of age with a history of ASCVD (hear and blood vessels diseases) or high-risk participants who have elevated bad cholesterol (LDL-C ≥1.8 mmol/L). The alternative model of care includes telephone support calls from a study nurse (after visits 1,2 and 4) and text messages to your mobile phone with healthy heart information.

The main question it aims to answer is to understand and compare an alternative model of care in comparison to the usual model of care by evaluating the study participants bad cholesterol values after 180 and 365 days of the study.

Each participant will take their medications as per usual care but may have the addition of Inclisiran, 284 mg 1.5 ml liquid in a single-use prefilled syringe for under skin administration. In accordance with the current medical practice guidelines for treating heart related conditions, Inclisiran and its product information will be made available for use in both care models.

All the participants who decide to take part in this study will be requested to do the following:

* Answer any questions from the study doctor or the study staff as accurately as possible when asked about changes in health status, medications, heart health, visits to other doctors or hospital admissions, planned surgery, even if they think none of these are related to the study.
* Study doctor will be able to inform them of which medications you can and cannot take as part of this study.
* To use mobile phone to receive text messages and/or questionnaires as proposed in the new model of care.
* Advise the study doctor if they plan to move away from the geographical area where the study is being conducted during the study period.
* Take the medications for cholesterol lowering treatment (such as a statin and/or ezetimibe) that are prescribed by the study doctor.
* Tell the study doctor or study staff as soon as possible about suspected participant / participant partner pregnancy.
* Tell the study doctor or study staff if they change their mind about taking part in the study.
* Attend all the visits (screening visit, visits 1, 2, 3, 4 and visit 5).
* Provide all the information that will enable the study team to contact them, i.e., inform the study staff if contact details change, provide contact details of a family member, etc.

DETAILED DESCRIPTION:
ASCVD remains a significant burden in the Australian population. Moreover, based on recent local data, it is clear that there are still opportunities to improve the management of this condition in Australia.

In collaboration with leading experts in the field, analysis of the gaps in management of cholesterol in Australia has been undertaken. Key areas identified include Lack of regular lipid testing in general practice, Limited access to full range of management tools, current therapies aren't achieving clinical guidelines and poor medication adherence.

To address these pain points, the ASCERTAIN study will implement a new model of care that has been co-created with leading cardiologists in Australia and feedback has been provided by a General Practitioner (GP) Advisory Committee.

As the primary purpose of this study is to assess the impact of a new model of care compared to usual care, Inclisiran and its approved Product Information will be made available in both arms to be used as per the treating physician's discretion. Participants taking part in this study will receive maximally tolerated statin and/or ezetimibe therapy with or without other LDL-C lowering therapies as per the treating physician's discretion.

The primary clinical question of interest is:

What is the effectiveness of a new model of care implementation strategy compared to usual care in patients who have not reached their LDL-target?

In the usual care arm:

1- The GPs will be educated on the European Society of Cardiology (ESC) guidelines and Guideline Directed Management therapy (GDMT)

In the new model of care arm:

1. The GPs will be educated on the ESC guidelines and Guideline Directed Management therapy (GDMT).
2. The Participants enrolled in this arm will be receiving monthly short message service (SMS) messages with regards to regarding cardiovascular health and appointment reminders (low touch engagement nudges).
3. In addition, Participants will receive telephone-based support calls from a study nurse trained in motivational interviewing. These telephone calls will cover diet, exercise, medication, and where necessary smoking cessation. A summary of any recommendations will then be sent to the primary care physician via email or letter. However, ultimately the primary care physician is responsible for the management of their patient.

The study will include male and female participants ≥18 years of age with a history of ASCVD (coronary heart disease, ischaemic cerebrovascular disease or peripheral arterial disease) or ASCVD-risk equivalents who have elevated LDL-C (≥1.8 mmol/L). A total of approximately 600 participants will be included in the study and will be randomised in a 1:1 ratio at approximately 20 sites across Australia.

For the purposes of defining the ASCVD-risk equivalent group, the Guidelines for the Management of Absolute Cardiovascular Disease Risk (2023) in Australian adults will be used. As per these guidelines, the online calculator www.cvdcheck.org.au (which is based on the Framingham Risk Equation) will be used to calculate an individual's estimated 5-year absolute CVD risk. High risk corresponds to >10% probability of CVD within the next 5 years.

Formal feasibility assessment will be completed by the Sponsor to ensure clinics are suitable for participation in the study.

Study sites may receive a list of patients who could qualify for the study. This list may be generated by a search of the practice database running a query for patients that satisfy the inclusion criteria. Alternatively, the sites may identify patients who could qualify for the study independently. The study sites will contact participants who meet the eligibility criteria.

Patient Reported Outcomes (PROs) will be completed by the participant electronically. Participants will receive a link to the questionnaire via text message or email.

The analysis will be performed at the end of the study, after the data for all participants are available. Unless otherwise specified, all statistical tests will be conducted against a two-sided alternative hypothesis, employing a significance level of 0.05.

Efficacy, safety, and other data will be summarised. For continuous variables, summary statistics (mean, standard deviation, median, interquartile range, minimum, and maximum) at each time point and for change from baseline to each time point will be reported by study arm. For discrete variables, frequency counts and percentages at each time point will be reported by study arm.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study
2. Males and females ≥18 years of age
3. Documented History of ASCVD

   a. Coronary heart disease (CHD):
   1. Prior myocardial infarction
   2. Prior coronary revascularisation (PCI or CABG)

   b. Cerebrovascular disease:
   1. Prior documented ischaemic stroke
   2. Documented Carotid artery stenosis >70%
   3. History of prior percutaneous or surgical carotid artery revascularisation.

   c. Peripheral arterial disease (PAD):
   1. History of prior percutaneous or surgical revascularisation of an iliac, femoral, or popliteal artery or aortic aneurysm in electronic patient history
   2. Prior surgical amputation of a lower extremity due to peripheral artery disease.

   OR ASCVD risk equivalents as per assessed by the online tool (>10% probability of CVD event within the next 5 years www.cvdcheck.org.au/calculator) or at clinically determined high risk.
4. Serum LDL-C above target ≥1.8 mmol/L (≥70 mg/dL) for ASCVD patients or ≥2.0 mmol/L for ASCVD risk equivalent patients
5. Not at Guideline directed cholesterol goals
6. On a stable dose of lipid-lowering therapy (such as a statin and/or ezetimibe) for ≥30 days before screening with no planned medication or dose change. Statin intolerant patients are eligible if intolerance is documented.

Exclusion Criteria:

1. Any medical or surgical history and or condition that might limit the individual's ability to take part in the study and/or put the participant at significant risk (according to physician's judgment).
2. Any underlying known disease, or surgical, physical, or medical condition that, in the opinion of the physician might interfere with the interpretation of the study results, including pregnancy.
3. Previous, current, or planned treatment with a monoclonal antibody targeting PCSK9.
4. Participants unable to access or unwilling to use mobile phone to receive text messages and/or questionnaires as proposed in the new model of care.
5. Participants who plan to move away from the geographical area where the study is being conducted during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Effect on LDL-C Concentration | Baseline and 180 Days
  LDL-C concentration at baseline and at day 180

SECONDARY OUTCOMES:
Effect on LDL-C Concentration | 365 Days
  LDL-C concentration at baseline and at day 365

OTHER OUTCOMES:
Patient satisfaction- Client Satisfaction Questionnaire | Baseline,180 and 365 Days
  CSQ-8 (Client Satisfaction Questionnaire) score at baseline, and days 180 and 365-Total scores range from. 8 to 32 with the higher number indicating greater satisfaction
Patient Activation Measure | Baseline,180 and 365 Days
  Patient activation measure (PAM) questionnaire score at baseline, and days 180 and 365 (Raw scores are transformed to a scaled of 0-100 ith higher PAM scores indicating higher patient activation)
LDL-C Concentration control | 90 and 270 Days
  Concentration of serum LDL-C to target (Primary prevention <2.0 mmol/L, Secondary prevention <1.8mmol/L, and secondary prevention for patients at very high risk <1.4mmol/L)
Blood Pressure Measure- Control over Risk factors | 90 and 270 Days
  Blood pressure value <130mmHg
HbA1c Value - Control over Risk factors | 90 and 270 Days
  HbA1c Value <7%
BMI Value - Control over Risk factors | 90 and 270 Days
  BMI <25kg/m2 (BMI is calculated by dividing the weight in Kilograms by the height in meters)
Medication adherence | 365 Days
  Proportion of patients reporting high levels of adherence to lipid lowering therapy between both arms.
Lowering absolute cardiovascular (CV) risk | 180 Days
  Absolute risk at day 180 as assessed by the CVD Check Calculator: www.cvdcheck.org.au/calculator).
Health care resourcing consumption | 180 and 365 Days
  The health care resourcing consumption of each of the models of care as assessed by Medicare item number utilisation if feasible.
Identify potential opportunities and challenges that can have an effect on scalability of the model of care for a broader population-1 | 180 and 365 Days
  Characterise study sites and their relationship to Intensification of LDL-C lowering therapy as per GDMT.
Identify potential opportunities and challenges that can have an effect on scalability of the model of care for a broader population-2 | 180 and 365 Days
  Characterise patients' demographics and their relationship to Intensification of LDL-C lowering therapy as per GDMT.
Identify potential opportunities and challenges that can have an effect on scalability of the model of care for a broader population-3 | 180 and 365 Days
  Characterise study sites and their relationship to effectiveness of CV risk factor lowering.
Identify potential opportunities and challenges that can have an effect on scalability of the model of care for a broader population-4 | 180 and 365 Days
  Characterise patients' demographics and their relationship to effectiveness of CV risk factor lowering.
Lp(a) levels | 180 Days
  Lp(a) levels at baseline and day 180
Changes in Lp(a) levels | 180 Days
  The percentage change in Lp(a) from baseline to Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholls, Principal Investigator — Monash University
Locations (1):
- Manningham General Practice, 200 High St, Templestowe Lower, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No